CLINICAL TRIAL: NCT01508273
Title: Development of an Aerobic and Resistance Training Feasibility Study for a Racially and Ethnically Diverse Sample of Breast Cancer Survivors
Brief Title: Lifestyle Intervention for High Risk Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-0743; K01CA158000 (NIH); NCI-2014-02453 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast Cancer Survivors; High risk cancer survivors; Stage II to IIIC breast cancer; African American; AA; Hispanic; Non-Hispanic White; Operable invasive breast carcinoma; Aerobic and resistance training; Pedometer; Telephone Counseling Calls; Physical activity report; PAR; Functional Assessment of Cancer Therapy-Breast; FACT-B; Health related quality of life; HRQOL
MeSH Terms: conditions — Breast Neoplasms | interventions — Resistance Training; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise Intervention Program Group (Experimental): At baseline study visit, participant shown how to complete the physical exercises performed while on study. Pedometer received to track physical activity. Resistance training bands given to use as part of the home-based exercise program. At the baseline study visit, directions received on how to use the study website. Access given to website that will allow tracking of exercise behavior and help set goals. Access given to an internet-based curriculum that will help teach about goal-setting, overcoming barriers to physical activity, self-management strategies, and time-management skills. Participant asked to visit website every week. Participant records activity and the number of steps taken every day on the website. Survey completed monthly about attitudes and beliefs about physical activity.
  Interventions: Behavioral: Exercise Program; Behavioral: Website; Behavioral: Survey
- Sedentary Behavior and Dietary Intervention Group (Other): Access given to internet-based curriculum to help teach about goal-setting, overcoming barriers to physical activity, self-management strategies, and time-management skills. Participants read information about improving the quality of their diet and cutting back on sedentary behavior. Participants record on the website how much television watched and how many fruits and vegetables eaten every day. Survey completed monthly about attitudes and beliefs about sedentary behavior and dietary intake.
  Interventions: Behavioral: Website; Behavioral: Survey
- Chair-based Study Group (Experimental): Patients participate in chair-based exercise study. Participants receive chair-based exercise DVD. Chair-based exercise program participation for a total of 8 weeks. Participants receive self-report assessments about quality of life and asked to participate in physical assessments of their balance and coordination.
  Interventions: Behavioral: Exercise DVD; Behavioral: Self-Report Assessments

INTERVENTIONS:
Behavioral: Exercise Program — Resistance training bands, guidebook, and pedometer given at baseline visit. Internet-based curriculum access given to teach goal-setting, overcoming barriers to physical activity, self-management strategies, and time-management skills. Access given website that will allow participant to track exercise behavior and help set goals.
  Arms: Exercise Intervention Program Group
Behavioral: Website — Website access given that allows participant to track exercise behavior and help to set goals.
  Arms: Exercise Intervention Program Group; Sedentary Behavior and Dietary Intervention Group
Behavioral: Exercise DVD — Participants receive chair-based exercise DVD. Participants in this chair-based exercise program for a total of 8 weeks.
  Arms: Chair-based Study Group
Behavioral: Survey — Exercise Intervention Program Group : Survey completion monthly about attitudes and beliefs about physical activity.
  Sedentary Behavior and Dietary Intervention Group: Survey completion monthly attitudes and beliefs about sedentary behavior and dietary intake.
  Arms: Exercise Intervention Program Group; Sedentary Behavior and Dietary Intervention Group
Behavioral: Self-Report Assessments — Self-report assessments given about quality of life and physical assessments of balance and coordination.
  Arms: Chair-based Study Group

SUMMARY:
The goal of this behavioral research study is to find out more about the health behaviors of cancer survivors. Researchers want to understand the cultural, social, and environmental factors related to physical activity and personal diet. Researchers also want to learn if cancer survivors who take part in lifestyle interventions have better overall health and quality of life than those who do not take part in these interventions.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will have a baseline study visit. This visit will include a physical exam, including measurements of your height and weight. Your hips, wrist, mid-arm, and waist will also be measured. You will also fill out questionnaires that contain items about your diet and exercise habits as well as questions about your quality of life.

Study Groups:

You will be randomly assigned (as in the flip of a coin) to 1 of 2 groups.

* Group 1 will take part in an exercise intervention program.
* Group 2 will take part in a sedentary behavior and dietary intervention group.

Group 1--Exercise Intervention:

At the baseline study visit, the study staff will show you how to complete the physical exercises you will perform while you are on study.

You will receive a pedometer that you can wear on your waistband to track your physical activity. The pedometer is the size of a deck of cards and will be worn throughout the study to track your progress.

You will be given resistance training bands to use as part of the home-based exercise program. At the baseline study visit, you will receive a directions on how to use the study website. In addition, the study coordinator will walk you through each of these exercises. After the study is complete, you will be allowed to keep the resistance training bands and pedometer.

Participants in Groups 1 will receive access to a website that will allow you to track your exercise behavior and help you set goals. This data will be recorded for you, and your progress will be graphed throughout the course of the study.

You will be given access to an internet-based curriculum that will help teach you about goal-setting, overcoming barriers to physical activity, self-management strategies, and time-management skills. You are being asked to visit the website every week to read that week's lesson materials and to set weekly goals. In addition to this weekly visits, you will need to record your activity and the number of steps you take every day on the website. Each month, you will be asked to fill our a survey about your attitudes and beliefs about physical activity.

Group 2--Parallel-Study Group:

Participants who are assigned to this group will received access to the same website as Group 1. You will also be asked to read information about improving the quality of your diet and cutting back on sedentary behavior ( for example, television viewing and overall sitting). The website will allow you to track your sitting and dietary behaviors and help you set goals. This data will be recorded for you, and your progress will be graphed throughout the course of the study.

Participants in Group 2 will be given access to curriculum that will help teach you about goal-setting, overcoming barriers to improving your diet and cutting back on sedentary behavior, as well as learn self-management strategies and time-management skills. You are being asked to visit the website once a week to read that week's lesson materials and to set weekly goals. In addition to this weekly visit, you will need to record on the website how much television you watch and how many fruits and vegetables you eat every day. Each month, you will be asked to fill our a survey about your attitude and beliefs about sedentary behavior and dietary intake.

6-Month Follow-up Visit: For both groups (Groups 1 & 2), at the 6-month follow-up visit, your weight and waist, hip, and arm measurements will be recorded and compared to your measurements from the baseline visit.

Length of Study:

For both groups, you will be taken off study if you experience side effects from taking part in the intervention, you are hospitalized for any reason, or you are diagnosed with a condition that needs a treatment not allowed while on this study.

Your participation on the study will be over once you have completed the 6-month visit.

This is an investigational study.

Up to 200 cancer survivors will take part in this study. Up to 150 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old at diagnosis
2. diagnosed with operable invasive cancer
3. have access to high speed internet
4. Phase 2 only: be currently sedentary (i.e., engage in < or = 60 minutes of purposeful moderate-intensity PA/week)
5. Phase 2 only: be overweight or obese (i.e., have a body mass index (BMI) > or = 25 kg/m^2)
6. speak English

Exclusion Criteria:

1. watch less than 3 hours of television per day
2. be currently enrolled in another intervention study or recently completed a study promoting healthy lifestyle behaviors (diet and/or exercise)
3. participants answering 'Yes' to one or more of the questions on the physical activity readiness questionnaire (PAR-Q) will need to obtain approval from a physician before they can participate in the intervention.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1150 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Health Behaviors of Breast Cancer Survivors | 6 months
  Data collected from mail-based surveys (n = 1,000) to assess intervention preferences, physical activity (PA), health related quality of life (HRQOL), and mediators of change (e.g., self-efficacy).

SECONDARY OUTCOMES:
Home-Based Exercise Feasibility | 6 months
  Rates of recruitment (% recruited out of the total number invited), retention (% completing the 6-month intervention), adherence (% completing 100% of study requirements), satisfaction, adverse events, and barriers to a home-based aerobic and resistance-training program.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Hajek, PHD, MS, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - The University of North Texas Health Science Center, Fort Worth, Texas
  - Memorial Herman Health Care System, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org